CLINICAL TRIAL: NCT02810925
Title: Weight Loss and Appetite Reduction and Their Correlation With Plasmatic Ghrelin Levels After Percutaneous Electrical Stimulation Dermatome T6 Associated With a Hypocaloric Diet
Brief Title: Weight Loss and Appetite Reduction After Percutaneous Electrical Stimulation Dermatome T6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Head of Neurostimulation Unit. Garcilaso Clinic, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ClinGarci 16-2
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PENS T6 and 1200 Kcal/day diet (Experimental): Patients undergo 12 sessions of percutaneous electrical stimulation of dermatome T6 (PENS T6), weekly, during 12 weeks. During this period they follow a hypocaloric 1200 Kcal/day diet.
  Interventions: Procedure: PENS T6; Dietary Supplement: Hypocaloric 1200 Kcal/day diet
- PENST6 + Normocaloric 2000 Kcal/day diet (Active Comparator): Patients undergo 12 sessions of percutaneous electrical stimulation of dermatome T6 (PENS T6), weekly, during 12 weeks. During this period they follow a normocaloric 2000 Kcal/day diet.
  Interventions: Procedure: PENS T6; Dietary Supplement: Normocaloric 2000 Kcal/day diet
- TENS T11/ T12 + 1200 Kcal/day diet (Placebo Comparator): Patients undergo 12 sessions of transcutaneous electrical stimulation of dermatomes T11-T12 , weekly, during 12 weeks. During this period they follow a hypocaloric 1200 Kcal/day diet.
  Interventions: Procedure: TENS T11/T12; Dietary Supplement: Hypocaloric 1200 Kcal/day diet
- 1200 Kcal/day diet (Active Comparator): Patients follow only a hypocaloric 1200 Kcal/day diet.
  Interventions: Dietary Supplement: Hypocaloric 1200 Kcal/day diet

INTERVENTIONS:
Procedure: PENS T6 — Patients undergo percutaneous electrical stimulation of dermatome T6, weekly, during 12 weeks.
  Arms: PENS T6 and 1200 Kcal/day diet; PENST6 + Normocaloric 2000 Kcal/day diet
Procedure: TENS T11/T12 — Patients undergo transcutaneous electrical stimulation of dermatomes T11-T12, weekly, during 12 weeks.
  Arms: TENS T11/ T12 + 1200 Kcal/day diet
Dietary Supplement: Hypocaloric 1200 Kcal/day diet — Patients follow a Hypocaloric 1200 Kcal/day diet during 12 weeks.
  Arms: 1200 Kcal/day diet; PENS T6 and 1200 Kcal/day diet; TENS T11/ T12 + 1200 Kcal/day diet
Dietary Supplement: Normocaloric 2000 Kcal/day diet — Patients follow a Normocaloric 2000 Kcal/day diet during 12 weeks.
  Arms: PENST6 + Normocaloric 2000 Kcal/day diet

SUMMARY:
The patients are randomized into 4 groups : Patients undergoing PENS of dermatome T6 in and a 1200 Kcal diet (Group 1), Patients undergoing PENS T6 and a 2000 Kcal/day, Patients undergoing transcutaneous electrical neurostimulation (TENS) of Dermatomes T11-T12 and following a 1200 Kcal diet and those patients following only a 1200 Kcal diet (Group 4). Weight loss, appetite and ghrelin levels at baseline and after treatment are investigated.

DETAILED DESCRIPTION:
The patients were randomized into 4 groups using an Internet randomization module: Patients undergoing PENS of dermatome T6 in conjunction with the implementation of a 1200 Kcal diet (Group 1), Patients undergoing PENS T6 and following a normocaloric diet (2000 Kcal/day) (Group 2), Patients undergoing transcutaneous electrical neurostimulation (TENS) of dermatomes in right iliac fossa (Dermatomes T11-T12) and following a hypocaloric diet (1200 Kcal/day) (Group 3) and those patients following only a 1200 Kcal diet (Group 4).

Weight loss, appetite and ghrelin levels, at baseline and after treatment, are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obesity (BMI>30 Kg/m2) or overweight (BMI 25-30 Kg/m2)

Exclusion Criteria:

* Untreated endocrine disease causing obesity
* Serious psychiatric illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | After 12 weeks of treatment
  Weight loss will be evaluated after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Castro, Study Chair — Clinica Garcilaso

IPD SHARING:
Plan to Share IPD: Yes
Data might be published in a journal, always preserving patients´ confidentiality.